CLINICAL TRIAL: NCT05502887
Title: The Endothelial Cell Dysfunction and Outcome Project for Hematological Neoplasms (EndoCDO-H). A Prospective Registry Study on Endothelial Functional Profile, Intervention Type and Clinical Outcome in Patients With Hematological Neoplasms
Brief Title: The Endothelial Cell Dysfunction and Outcome Project for Hematological Neoplasms
Acronym: EndoCDO-H
Status: Recruiting | Type: Observational
Sponsor: Prof. Dr. Thomas Luft (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Thomas Luft, Professor, University Hospital Heidelberg
Organization: University Hospital Heidelberg (Other)
Other Study IDs: EndoCDO-H
Record Dates: First submitted 2022-06-09; First posted 2022-08-16 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Hematological Neoplasm; Endothelial Dysfunction
Keywords: endothelial cells; biomarkers; endothelial activation and stress index (EASIX); endothelial complications; non-relapse mortality; in vivo microscopy
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and bone marrow samples, plasma and serum including liquid biopsies (cfDNA) are collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Researched Group: All patients with newly diagnosed or preexistent hematological neoplasms at participating centers are intended to be registered within EndoCDO-H. Prior to inclusion, patients have to give their written informed consent.
  Interventions: Diagnostic Test: Sublingual in vivo microscopy with the Glycocheck microscope

INTERVENTIONS:
Diagnostic Test: Sublingual in vivo microscopy with the Glycocheck microscope — For the collection of longitudinal microscopy data, sublingual in vivo microscopy with the Glycocheck microscope will be performed at the following timepoints: 2-3 x between day (D) -28 of allogeneic HSCT or CAR T cell therapy and before start of the conditioning regimen, once between D2-D14, once between D15-28, once between D30- D100 and at the onset of endothelial complications such as acute GvHD, TMA, sepsis, VOD and IPS following allogeneic HSCT or CAR T cell therapy. Sublingual microscopy requires 15-30 minutes and is similar to sublingual temperature measurement. To this extent, a tube with a diameter of approximately 1cm carrying a microscope at the tip is inserted into the mouth and under the tongue to measure endothelial structures (blood flow through small capillaries). Biological samples are collected and processed within the established Biobank of the Internal Medicine V of the Heidelberg University Hospital.

SUMMARY:
The endothelium is a semipermeable monolayer of endothelial cells (EC) organized as a complex biological interface that separates all tissues from circulating blood. Any anti-neoplastic or immune therapy will directly challenge the endothelial layer, with a substantial risk of damaging EC or exacerbating pre-existing endothelial cell dysfunction.

In our previous researchs the concepts of "endothelial vulnerability" and "endothelial cell dysfunction" for initial diagnosis of patients with hematological disorders, e.g. myelodysplastic syndromes as well as COVID-19 patients were designed. The novel and pre-existing endothelial vulnerability markers and markers of endothelial cell dysfunction or damage such as endothelial activation and stress index (EASIX) were also defined, validated and their prognostic role for treatment-related mortality and for a variety of allo- and CART-specific endothelial complications were established. However, the exact relationship of EASIX and other markers with endothelial cell biology are not known and require further clarification.

Primary aims are to demonstrate that EASIX represents a systemic response of the organism to local or systemic loss of endothelial glycocalyx as visualized by sublingual microscopy and to establish EASIX, biomarkers and in vivo microscopy of sublingual and (in perspective) recto-sigmoidal capillary beds as prognostic markers of response to anti-neoplastic therapy, treatment-related toxicity and mortality (TRM) and overall survival (OS). Secondary objectives include the creation of a comprehensive database with information on endothelial, clinical, pathological and molecular characteristics of patients with hematological malignancies as well as the establishment of a repository of biospecimens for endothelial marker analyses from patients with hematological malignancies.

We hypothesize that reduced endothelial glycocalyx thickness will permit direct interactions of leukocytes and platelets with endothelial cells, resulting in cellular activation (increased LDH), loss of platelets due to activation and microembolism, and ensuing kidney damage. As a first prospective analysis, we will answer the question if EASIX and serum endothelial biomarkers correlate with sublingual glycocalyx thickness, and if these parameters combine to predict outcome after anti-neoplastic therapy including alloSCT and CART.

DETAILED DESCRIPTION:
Functional heterogeneity is a hallmark of the endothelial cell system. The hypothetical functional definition of ECs as input-output devices emphasizes their role as direct responders to a variety of challenges such as blood pressure, temperature, pH and oxygen pressure, and serum factors. Maintaining homeostasis of tissue perfusion is an important function of ECs that are continuously exposed to stimuli provided by the alternative complement pathway, coagulation factors, cytokines, activated platelets, leukocytes, and occasional infectious agents. Due to their distribution over space and time, hardly two ECs will be exposed to the same set of input signals 8. Moreover, stochastic or inheritable heterogeneous DNA methylation patterns add to the functional variability of seemingly "homogeneous" mature EC populations. Therefore, tissue-specific stress responses of ECs can explain that even during systemic EC dysfunction (e.g. due to calcineurin inhibitors, viruses, TBI etc.), microangiopathy develops locally in individual patients. This functional heterogeneity has to be considered in all attempts to define clinical diagnostic criteria for endothelial complications after hematological anti-neoplastic therapy including alloSCT and CART infusions.

Over the last years, our group has developed the concepts of "endothelial vulnerability" and "endothelial cell dysfunction" that pre-exist before alloSCT and CART infusions and at initial diagnosis of patients with hematological disorders, e.g. myelodysplastic syndromes, but also in COVID-19 patients. We have defined and validated novel and pre-existing endothelial vulnerability markers (e.g. single nucleotide polymorphisms in THBD (Thrombomodulin) and CD40 Ligand; serum levels of Angiopoietin-2, serum nitrates, asymmetric dimethyl-arginine (ADMA), testosterone deficiency, interleukin-18), and markers of endothelial cell dysfunction or damage (e.g. suppressor of tumorigenicity (ST)-2, interleukin-18, insulin-like growth factor 1 (IGF1), CXCL8), and we have established their role as prognostic markers for treatment-related mortality and for a variety of allo- and CART-specific endothelial complications.

The heterogeneity of EC explains why global one-for-all markers were not found within the group of endothelial-derived and endothelial-specific prognostic factors. We therefore developed the Endothelial activation and stress index, EASIX, as a marker that represents the response of the organism to endothelial dysfunction. EASIX represents an interplay of the basic laboratory parameters (LDH*creatinine/platelets) observed at onset of the most severe endothelial complication after alloSCT, i.e. transplant-associated thrombotic microangiopathy (TAM). EASIX correlated with endothelial serum markers such as IL18, ANG2 and IGF1 and predicted outcome in a variety of clinical settings including COVID-19. However, the exact relationship of EASIX to endothelial cell biology requires further clarification. We hypothesize that reduced endothelial glycocalyx thickness will permit direct interactions of leukocytes and platelets with endothelial cells, resulting in cellular activation (increased LDH), loss of platelets due to activation and microembolism, and ensuing kidney damage.

Thus, key areas of interest are:

* Comprehensive collection and intercorrelation of endothelial parameters before, during and after new lines of therapy including in vivo microscopy, ECHO cardiography, EASIX, body weight, endothelial serum markers including, but not restricted to, ST2, ANG2, IL18, IL8, sCD141, Hyaluronan, Syndecan-1, CXCL9, Leptin, Adiponectin, Testosterone, and others.
* Correlation of EASIX with glycocalyx thickness and capillary flow measured by in vivo microscopy of the capillary bed.
* Systematic collection of clinical data on known endothelial complications, including, but not restricted to, sepsis, septic shock, macrophage activation syndrome, veno-occlusive disease / sinusoidal obstruction syndrome (SOS/VOD), thrombotic microangiopathy, idiopathic pneumonia syndromes (IPS), paraneoplastic syndromes, engraftment syndrome, persistent intestinal inflammation, cachexia, and others.
* Systematic collection and evaluation of comprehensive biological specimens and information from patients with hematological neoplasms, including data on the genomic, transcriptomic, epigenomic and proteomic "landscapes" as well as expression of surface antigens of hematological disease subtypes, to identify novel prognostic and predictive endothelial parameters as well as entry points for targeted therapeutic interventions that protect the endothelium.
* Multivariable prediction analyses of endothelial parameters on outcome and endothelial complications.

The above challenges are ideally met by a registry study with a sufficient population size to answer relevant questions in rare therapy-related complications and rare cancer entities.

The aim is to set up a registry study that covers systematic and comprehensive clinical data acquisition, and longitudinal banking of serum, blood cells and bone marrow samples of patients with hematological diseases, with focus on in vivo microscopy, EASIX, and serum endothelial markers.

This resource will spur patient-oriented investigations into relationships between endothelial, clinical and tumor-biological parameters in hematological neoplasms and lay the groundwork for novel, supportive treatment approaches protecting the endothelial system in poorly understood and difficult-to-treat subsets.

As a first prospective analysis, we will answer the question if EASIX and serum endothelial biomarkers correlate with sublingual glycocalyx thickness, and if these parameters combine to predict outcome after anti-neoplastic therapy including alloSCT and CART.

ELIGIBILITY:
Inclusion Criteria:

* Suspected or proven diagnosis of hematological neoplasms according to the WHO Classification of Tumours of Haematopoietic and Lymphoid Tissues;
* Age ≥18 years;
* Ability to understand nature and individual consequences of the registry;
* Written informed consent;
* Subjects who are physically or mentally capable of giving consen.

Exclusion Criteria:

- Severe neurological or psychiatric disorder interfering with the ability to give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with newly diagnosed or preexistent hematological neoplasms at participating centers are intended to be registered within EndoCDO-H. Prior to inclusion, patients have to give their written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2027-06-07 (Estimated); Study Completion 2032-06-07 (Estimated)

PRIMARY OUTCOMES:
overall survival | observation peroid 10 years
  Time period between date of informed consent to alive at last follow-up or death

SECONDARY OUTCOMES:
side effects | observation peroid 10 years
  toxicity measured according to CTC AE version 5.0
Treatment adaptation | observation peroid 10 years
  reduction of dose intensity
endothelial glycocalyx | observation peroid 10 years
  endothelial glycocalyx measured by sublingual microscopy

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Thomas Luft, Principal Investigator — Heidelberg University
Locations (1):
- Department of Internal Medicine V, Heidelberg University Hospital, Heidelberg, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Luft T, Dreger P, Radujkovic A. Endothelial cell dysfunction: a key determinant for the outcome of allogeneic stem cell transplantation. Bone Marrow Transplant. 2021 Oct;56(10):2326-2335. doi: 10.1038/s41409-021-01390-y. Epub 2021 Jul 12. PMID 34253879
- [Background] Luft T, Wendtner CM, Kosely F, Radujkovic A, Benner A, Korell F, Kihm L, Bauer MF, Dreger P, Merle U. EASIX for Prediction of Outcome in Hospitalized SARS-CoV-2 Infected Patients. Front Immunol. 2021 Jun 23;12:634416. doi: 10.3389/fimmu.2021.634416. eCollection 2021. PMID 34248931
- [Background] Luft T, Benner A, Jodele S, Dandoy CE, Storb R, Gooley T, Sandmaier BM, Becker N, Radujkovic A, Dreger P, Penack O. EASIX in patients with acute graft-versus-host disease: a retrospective cohort analysis. Lancet Haematol. 2017 Sep;4(9):e414-e423. doi: 10.1016/S2352-3026(17)30108-4. Epub 2017 Jul 18. PMID 28733186
- [Background] Luft T, Benner A, Terzer T, Jodele S, Dandoy CE, Storb R, Kordelas L, Beelen D, Gooley T, Sandmaier BM, Sorror M, Zeisbrich M, Radujkovic A, Dreger P, Penack O. EASIX and mortality after allogeneic stem cell transplantation. Bone Marrow Transplant. 2020 Mar;55(3):553-561. doi: 10.1038/s41409-019-0703-1. Epub 2019 Sep 26. PMID 31558788
- [Derived] Simons L, Alasfar L, Qadoura M, Buhl J, Sunderer F, Korell F, Ikonomidis I, Dietrich M, Seidlitz S, Vink H, Maier-Hein L, Schmitt M, Schlenk RF, Carsten Muller-Tidow, Dreger P, Luft T. Comprehensive assessment of endothelial dysfunction before cellular therapy: EASIX, local imaging, and systemic biomarkers. Blood Vessel Thromb Hemost. 2025 Sep 10;2(4):100105. doi: 10.1016/j.bvth.2025.100105. eCollection 2025 Nov. PMID 41334245